CLINICAL TRIAL: NCT06457529
Title: The Effect of Dry Needling and Prolotherapy on Pain, Function, and Quality of Life in Patients With Cervical Radiculopathy.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/721
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional treatment with Prolotherapy (Experimental)
  Interventions: Diagnostic Test: conventional treatment with Prolotherapy
- Dry Needling and conventional treatment (Other)
  Interventions: Other: Dry Needling and conventional treatment

INTERVENTIONS:
Diagnostic Test: conventional treatment with Prolotherapy — Group A got prolotherapy along with conven¬tional treatment, which includes ultrasonic therapy for 10 minutes. The intensity will be 3MHz at 1.0 watts/cm2.
  Prolotherapy is an injection treatment used to relieve pain. Your healthcare provider will inject a small amount of an irritant into your body. Dextrose (sugar) solution is the most commonly injected irritant. Proponents of prolotherapy claim it relieves pain by jumpstarting your body's natural healing abilities.
  Arms: conventional treatment with Prolotherapy
Other: Dry Needling and conventional treatment — Group B Subjects in Group B will get Dry Needling along with conventional treatment, which includes ultrasonic therapy for 10 minutes. The intensity will be 3MHz at 1.0 watts/cm2.
  Trigger-point dry needling is an invasive procedure where a fine needle or acupuncture needle is inserted into the skin and muscle
  Arms: Dry Needling and conventional treatment

SUMMARY:
Cervical radiculopathy is characterized by neurological dysfunction caused by compression and inflammation of the spinal nerves or nerve roots of the cervical spine. Rolotherapy is a regenerative therapeutic method that consists of injecting irritant solutions into the injured areas.

DETAILED DESCRIPTION:
Hyperosmolar dextrose is the most common agent. Administering proliferant substances can accelerate the tissue healing process by inducing cellular rupture and inflammatory response, leading to collagen deposition, cellular growth factor production, and regeneration. Dry needling used to relieve trigger point release in deep and superficial muscles. Both treatment interventions will apply to cervical radiculopathy patients to measure the effectiveness of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 20-50 years
* Both male and female
* Unilateral pain starting in the cervical spine and radiating to the upper limb.
* Pain aggravated by upper limb movement
* Restricted range of motion of arm

Exclusion Criteria:

* History of Spinal infection
* Spinal Cord Injury
* History of Vertebral tumor and factures
* History of cervical or intracranial surgery
* History of Radiating pain to bilateral upper limb.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | 12 Months
  The NDI has become a standard instrument for measuring self-rated disability due to neck pain and is used by both clinicians and researchers. Each of the 10 items scores from 0 to 5. The maximum score is 50. The obtained score can be multiplied by two to produce a percentage score
WHO Quality of Life | 12 months
  The QOLS is a reliable and valid instrument for measuring quality of life from the perspective of the patient. It focuses on domains that come from the qualitative descriptions of a wide range of adults across gender, cultural and language groups.Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale (16, 17). The physical health domain includes items on mobility, daily activities, functional capacity, energy, pain, and sleep

CONTACTS AND LOCATIONS:
Locations (1):
- Iqbal Mahmooda Hospital, Iffat Anwar Medical Complex and Life line Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No